CLINICAL TRIAL: NCT03206450
Title: Effects of Modern Chemotherapy Regimens on Spermatogenesis and Steroidogenesis in Adolescent and Young Adult (AYA) Survivors of Osteosarcoma
Brief Title: Biospecimen Analysis in Determining Effects of Chemotherapy on Fertility in Osteosarcoma Survivors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALTE16C1; NCI-2017-01152 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE16C1 (Other: Children's Oncology Group); COG-ALTE16C1 (Other: DCP); ALTE16C1 (Other: CTEP); R01CA175216 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — saliva, semen, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen collection): Participants complete a health questionnaire over 30-45 minutes. Patients also provide saliva and semen samples and undergo collection of blood.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and provide saliva and semen samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies saliva, semen, and blood samples to determine effects of chemotherapy on fertility in osteosarcoma survivors. Study biospecimen samples from osteosarcoma survivors in the laboratory may help doctors learn whether chemotherapy causes fertility problems and to learn more about the long term effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether infertility and/or biomarkers of spermatogenesis and steroidogenesis differ in male osteosarcoma survivors treated with cisplatin with or without ifosfamide compared to male controls without a history of cancer.

II. Evaluate whether cisplatin with or without ifosfamide for the treatment of osteosarcoma alters sperm deoxyribonucleic acid (DNA) methylation.

EXPLORATORY OBJECTIVES:

I. Evaluate the role of genetic susceptibility in the development of impairments in spermatogenesis or steroidogenesis with contemporary regimens for the treatment of osteosarcoma.

OUTLINE:

Participants complete a health questionnaire over 30-45 minutes. Patients also provide saliva and semen samples and undergo collection of blood.

ELIGIBILITY:
Inclusion Criteria:

* Received upfront therapies for osteosarcoma, which included cisplatin, (with or without other agents)
* Patient must have completed cancer treatment >= 2 years prior to study enrollment
* Osteosarcoma survivors without a systemically treated relapse or subsequent malignancy

  * Note: History of relapse or second malignancy is permitted if treated with local therapy only (e.g. surgery, radiation)
* Able to speak, read and write in English, French or Spanish
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Osteosarcoma survivors who receive upfront therapies for osteosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Infertility | Up to 4 years
  The American Society of Reproductive Medicine's definition of "infertility" as "… the failure to achieve a successful pregnancy after 12 months or more of regular unprotected intercourse" will be used to categorize patients as to a history of infertility. Based on interview questions regarding each subject's personal and partner's history of medical investigations and treatment for infertility, an attempt will be made to further distinguish each subject's history of infertility as being due to the male (study subject), the female or indeterminate. Will determine whether infertility differ in male osteosarcoma survivors treated with cisplatin with or without ifosfamide compared to male controls without a history of cancer. Will be analyzed using unconditional logistic regression models to estimate odds ratios and 95% confidence intervals for the associations of chemotherapy group with abnormal values as defined in clinical practice.
Follicle stimulating hormone levels | Up to 4 years
  Will be measured by immunofluorometric assay. Will be analyzed using unconditional logistic regression models to estimate odds ratios and 95% confidence intervals for the associations of chemotherapy group with abnormal values as defined in clinical practice.
Luteinizing hormone levels | Up to 4 years
  Will be measured by immunofluorometric assay. Will be analyzed using unconditional logistic regression models to estimate odds ratios and 95% confidence intervals for the associations of chemotherapy group with abnormal values as defined in clinical practice.
Testosterone levels | Up to 4 years
  Will be measured by radioimmunoassay. Will be analyzed using unconditional logistic regression models to estimate odds ratios and 95% confidence intervals for the associations of chemotherapy group with abnormal values as defined in clinical practice.
Serum inhibin B | Up to 4 years
  Will be measured by enzyme-linked immunosorbent assay. Will be analyzed using unconditional logistic regression models to estimate odds ratios and 95% confidence intervals for the associations of chemotherapy group with abnormal values as defined in clinical practice.
Sperm concentration | Up to 4 years
  Sperm concentration (per mL) will be assessed by Computer Assisted Sperm Analysis. Three separate counts will be performed and the results averaged. Will be analyzed using unconditional logistic regression models to estimate odds ratios and 95% confidence intervals for the associations of chemotherapy group with abnormal values as defined in clinical practice.
Sperm morphology | Up to 4 years
  Sperm morphology will be assessed. Will be analyzed using unconditional logistic regression models to estimate odds ratios and 95% confidence intervals for the associations of chemotherapy group with abnormal values as defined in clinical practice.
Sperm deoxyribonucleic acid methylation | Up to 4 years
  Genome-wide differentially methylated regions will be identified using methylated deoxyribonucleic acid immunoprecipitation followed by next generation sequencing analysis methylated deoxyribonucleic acid immunoprecipitation sequencing using pooled deoxyribonucleic acid. Sperm deoxyribonucleic acid differentially methylated regions will be confirmed in the pooled samples by bisulfite treatment of genomic deoxyribonucleic acid to convert cytosine to thymine followed by next generation sequencing for a bisulfite-sequencing analysis. Thus, methylated deoxyribonucleic acid immunoprecipitation- sequencing is used to identify the differentially methylated regions and bisulfite sequencing used to confirm the differentially methylated regions at the CpG level resolution. Pyrosequencing will be used involving next generation sequencing after polymerase chain reaction of individual sperm deoxyribonucleic acid samples to assess individual differentially methylated regions.

OTHER OUTCOMES:
Role of genetic susceptibility in the development of impairments in spermatogenesis or steroidogenesis with contemporary regimens for the treatment of osteosarcoma | Up to 4 years
  Analysis will be descriptive in nature and will be used to generate hypotheses for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Margarett Shnorhavorian, Principal Investigator — Children's Oncology Group
Locations (99):
- United States (93):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan